CLINICAL TRIAL: NCT05298020
Title: A Single-arm Phase II Study of Envafolimab Combined With Endostar and Nab-paclitaxel Plus Gemcitabine for First-line Treatment of Advanced Pancreatic Cancer
Brief Title: Envafolimab Combined With Endostar and Chemotherapy for First-line Treatment of Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2022-ENVA001
Record Dates: First submitted 2022-03-18; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Advanced Pancreatic Cancer
Keywords: Advanced pancreatic cancer; Envafolimab; Endostar; AG regimen
MeSH Terms: interventions — envafolimab; Immunotherapy; endostar protein; Endostatins; Taxes; Drug Therapy; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab and Endostar plus AG regimen (Experimental): Envafolimab:400mg,sc,d1,Q4W; Endostar：210mg，CIV72h，d1-3，Q4W； Chemotherapy:AG (nab-paclitaxel:125mg/m2,iv,d1,d8,Q4W；gemcitabine：1000mg/m2, iv,d1,d8，Q4W).
  Interventions: Drug: Envafolimab; Drug: Endostar; Drug: Nab paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Envafolimab — 400mg,sc,d1,Q4W
  Other Names: Immunotherapy
Drug: Endostar — 210mg，CIV72h，d1-3，Q4W
  Other Names: endostatin
Drug: Nab paclitaxel — 125mg/m2,iv,d1,d8,Q4W
  Other Names: Chemotherapy
Drug: Gemcitabine — 1000mg/m2, iv,d1,d8，Q4W
  Other Names: Chemotherapy

SUMMARY:
This is a single-arm, open-label, exploratory study to evaluate efficacy and safety of envafolimab combined with endostar and nab-paclitaxel plus gemcitabine for first-line treatment of advanced pancreatic cancer.

DETAILED DESCRIPTION:
This study is a prospective, open-label, single-arm, exploratory clinical study.

Recruited 20 subjects who met the inclusion criteria and received Endostar+Envofolimab+Nab-paclitaxel/Gemcitabine (AG regimen) chemotherapy according to the study plan. Treatment duration and dose can be adjusted according to patient tolerance until disease progression or intolerable toxicity, or other conditions determined by the investigator. During the trial, the efficacy indicators and safety indicators were observed.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven pancreatic cancer ；
* Age ≥ 18 years old, gender is not limited ； Expected survival ≥ 3 months ； ECOG 0-1； At least one measurable objective tumor lesion by spiral CT examination, the maximum diameter ≥ 1cm（according to RECIST 1.1）； No previous chemotherapy, radiotherapy, immunotherapy, targeted therapy； The function of major organs is good, that is, the relevant inspection indicators within 14 days before enrollment meet the following requirements：（Hemoglobin ≥ 90 g/L (no blood transfusion within 14 days);Neutrophil count > 1.5×109/L; Platelet count ≥ 100×109/L;Total bilirubin ≤ 1.5×ULN (upper limit of normal);Blood alanine aminotransferase (ALT) or blood aspartate aminotransferase (AST) ≤2.5×ULN; if liver metastases, ALT or AST ≤ 5×ULN;Endogenous creatinine clearance ≥ 60 ml/min (Cockcroft-Gault formula);Cardiac Doppler Ultrasound Assessment: Left Ventricular Ejection Fraction (LVEF) ≥ 50% ）；

Exclusion Criteria:

* Patients with other malignant tumors in the past or at the same time, and those tumors that are judged by the investigator to not affect the patient's life in the short term can be excluded； Participated in clinical trials of other drugs within four weeks ； Patients with known CNS metastases or a history of CNS metastases prior to screening. For patients with clinically suspected central nervous system metastasis, CT or MRI examination must be performed within 28 days before enrollment to exclude central nervous system metastasis; Patients with a history of unstable angina pectoris; newly diagnosed angina pectoris within 3 months before screening or myocardial infarction events within 6 months before screening; arrhythmia (including QTcF: male ≥ 450 ms, female ≥ 470 ms) requires Long-term use of antiarrhythmic drugs and New York Heart Association class ≥ II cardiac insufficiency; Urine routine indicates urine protein ≥++ and confirmed 24-hour urine protein quantification >1.0 g; For female subjects: should be surgically sterilized, postmenopausal, or agree to use a medically approved contraceptive during the study treatment period and within 6 months after the end of the study treatment period; Serum or urine pregnancy test must be negative within 7 days and must be non-nursing. Male subjects: should be surgically sterilized, or agree to use a medically approved contraceptive during the study treatment period and within 6 months after the end of the study treatment period; Have used immune targeted therapy drugs; Have a history of immunodeficiency, or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation; Infectious pneumonia, non-infectious pneumonia, interstitial pneumonia and other patients who need corticosteroids; History of chronic autoimmune diseases, such as systemic lupus erythematosus; history of inflammatory bowel disease such as ulcerative colitis, Crohn's disease, history of chronic diarrheal diseases such as irritable bowel syndrome; history of sarcoidosis Medical history or history of tuberculosis; history of active hepatitis B, hepatitis C and HIV infection; Patients with allergic reactions to human or camel-derived monoclonal antibodies; Those who have a history of psychotropic substance abuse and cannot quit or have mental disorders; Pleural effusion or ascites with clinical symptoms requiring clinical intervention; According to the judgment of the investigator, there are concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 months
  Objective response rate
PFS | 6 months
  Progressives free survival

SECONDARY OUTCOMES:
OS | 12 months
  Overall survival
DCR | 12 months
  disease controll rate
AEs | 12 months
  Percentage of participants experiencing grade 3-5 adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No